CLINICAL TRIAL: NCT03014921
Title: Effet de l'Injection de Fer Sur la Donation Sanguine, étude randomisée et contrôlée
Brief Title: Impact of Iron Injection on Blood Donation
Acronym: FERDOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nicolas Leuenberger (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Sponsor-Investigator, Nicolas Leuenberger, PhD, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2016-00324
Record Dates: First submitted 2016-12-23; First posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Iron Deficiency
MeSH Terms: conditions — Iron Deficiencies | interventions — Iron; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo injection group (Placebo Comparator): saline solution injection as placebo
  Interventions: Other: saline solution injection
- iron injection group (Active Comparator): iron injection
  Interventions: Other: iron injection

INTERVENTIONS:
Other: iron injection — Injection of a 250mL saline solution added with 500mg of iron (Ferinject)
  Arms: iron injection group
Other: saline solution injection — Injection of a 250mL saline solution
  Arms: placebo injection group

SUMMARY:
This trial study and compare in blood and urinary matrices the impact of an iron injection on proteins involved in iron metabolism during a blood donation. The goal is to study the impact of an iron injection on detection markers of a blood donation in the anti-doping field

DETAILED DESCRIPTION:
This study aim to investigate the impact of an iron injection on the proteins involved in iron metabolism during blood donation and to compare the blood and urinary matrix. A messenger RNA profiling will be performed as well. The goal is to investigate the impact of iron injection on the markers of blood donation detection in the anti-doping field.

The study will take place over a period of 8 weeks.

Volunteers will be randomly assigned to two groups. Randomization will be provided by a software made for this purpose. An injection of 500 mg of iron in 250mL of saline solution or a placebo injection containing only the saline solution will be performed. Standard blood sampling (in the arm) and finger prick blood sampling will be carried out. After that, 500 mL blood donation will be done. Standard blood sampling and finger prick blood sampling will be performed before and after the donation.

The study will be done in "simple blind", meaning that volunteers will not know if they get iron or saline solution.

On the days of iron or saline solution injection and blood donation, blood sampling will be done up to 12 hours after the injection. After that, blood sampling will be scheduled up to 30 days after blood donation at a rate of once a day (except for the weekends).

ELIGIBILITY:
Inclusion Criteria:

* Male between 20 and 35 yo
* BMI between 18 and 30
* Ferritin < 50ug/l
* Transferrin saturation < 20 if ferritin between 20 and 50ug/l

Exclusion Criteria:

* high level athlete
* blood donation within 6 months before the study
* liver disorder

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2016-12; Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Serum ferritin level variations due to iron injection or blood donation | 8 weeks
  measurements will be done in ug/l

SECONDARY OUTCOMES:
Hemoglobin level variations due to iron injection or blood donation | 8 weeks
  measurements will be done in g/dL
Reticulocyte% variations due to iron injection or blood donation | 8 weeks
  measurements will be done in %

IPD SHARING:
Plan to Share IPD: No